CLINICAL TRIAL: NCT01802268
Title: Outcomes of Planned Conversion From Tacrolimus to Sirolimus-based Immunosuppressive Regimen in de Novo Kidney Transplant Recipients
Brief Title: Planned Conversion From TAC to SRL-based Regimen in de Novo Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helio Tedesco Silva Junior (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Helio Tedesco Silva Junior, PhD, Hospital do Rim e Hipertensão
Organization: Hospital do Rim e Hipertensão (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E8-3328
Record Dates: First submitted 2013-02-22; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Transplant
Keywords: sirolimus; tacrolimus; early conversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Active Comparator): Conversion from Tacrolimus to Sirolimus
  Interventions: Drug: Conversion from Tacrolimus to Sirolimus
- Tacrolimus (Active Comparator): Maintenance on tacrolimus
  Interventions: Drug: Maintenance on tacrolimus

INTERVENTIONS:
Drug: Conversion from Tacrolimus to Sirolimus
  Arms: Sirolimus
Drug: Maintenance on tacrolimus
  Arms: Tacrolimus

SUMMARY:
Background Early conversion from calcineurin inhibitor to mammalian target of rapamycin inhibitor is one of the immunosuppressive strategies that have been investigated to mitigate long-term CNi associated adverse events. This study aims to evaluate the conversion from tacrolimus to sirolimus in de novo kidney transplant recipients.

This multicenter, open-label study, planned to enroll 297 patients initially treated with tacrolimus, enteric-coated mycophenolate sodium (1440 mg/day, orally) and prednisone. The primary objective is to show superior glomerular filtration rate in the SRL group at 24 months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years,
* recipients of first kidney transplant from brain dead deceased or living related non-HLA identical donors not older than 65 years,
* patients had to receive an ABO compatible organ with a CDC negative crossmatch and a peak panel reactive antibody lower that 30%,
* all patients agreed to use contraceptive methods during the study and up to 3 months after study drug discontinuation.

Exclusion Criteria:

* patients with chronic kidney diseases due to focal and segmental glomerulosclerosis and membranoproliferative glomerulonephritis,
* patients with active infection or positive for hepatitis B or C or human immunodeficiency viruses,
* patients with previous history of malignancy,
* patients with significant hematological or metabolic laboratorial abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2008-02; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Renal Function calculated using the 4 variable MDRD formula | 24 months

SECONDARY OUTCOMES:
Survival free from first treated biopsy confirmed acute rejection episodes (tBCAR) > IA according to Banff 1997 classification. | 24 months
Incidence of all treated acute rejections. | 24 months
Incidence and severity of all tBCAR. | 24 months
Patient and graft survival. | 24 months
Incidence of treatment discontinuation | 24 months
Incidence of adverse events. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Helio T. Silva Junior, PhD, Principal Investigator — Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil; Claudia R. Felipe, PhD, Study Chair — Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil; Valter D. Garcia, PhD, Study Chair — Kidney & Pancreas Transplant Unit, Santa Casa de Misericordia, Porto Alegre, Brazil; Elias D. Neto, PhD, Study Chair — Renal Transplant Service, Hospital das Clínicas, University of São Paulo School of Medicine, São Paulo, Brazil; Mario A. Filho, PhD, Study Chair — Instituto de Urologia e Nefrologia & Medical School-FAMERP/HB-FUNFARME, São José do Rio Preto-SP, Brazil; Fabiana LC Cortieri, PhD, Study Chair — Hospital University Evangélico de Curitiba, Curitiba, Parana, Brazil; Deise BM Carvalho, PhD, Study Chair — Nephrology Service, Bonsucesso General Hospital. Rio de Janeiro, Brazil; Jose OM Pestana, PhD, Study Director — Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil
Locations (6):
- Brazil (6):
  - Hospital University Evangélico de Curitiba, Curitiba, Parana, Brazil, Curitiba, Paraná
  - Nephrology Service, Bonsucesso General Hospital. Rio de Janeiro, Brazil, Rio de Janeiro, Rio de Janeiro
  - Kidney & Pancreas Transplant Unit, Santa Casa de Misericordia, Porto Alegre, Brazil, Porto Alegre, Rio Grande do Sul
  - Instituto de Urologia e Nefrologia & Medical School-FAMERP/HB-FUNFARME, São José do Rio Preto-SP, Brazil, São Jose Do Rio Preto, São Paulo
  - Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil, São Paulo, São Paulo
  - Renal Transplant Service, Hospital das Clínicas, University of São Paulo School of Medicine, São Paulo, Brazil., São Paulo, São Paulo